CLINICAL TRIAL: NCT03167034
Title: Effect of Acetazolamide on Right Ventricular Function During Exercise in Patients With Chronic Obstructive Pulmonary Disease at Altitude. A Randomized, Placebo-controlled, Double-blind Parallel Trial.
Brief Title: Effect of Acetazolamide on Right Ventricular Function During Exercise in Patients With Respiratory Disease at Altitude
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-00137F
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exercise; echocardiography; right ventricular function; obstructive airway disease; emphysema; acetazolamide; altitude
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Lung Diseases, Obstructive; Emphysema | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACETAZOLAMIDE oral capsule (Active Comparator): Acetazolamide 375mg/day (capsule @125 mg: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m
  Interventions: Drug: ACETAZOLAMIDE oral capsule
- PLACEBO oral capsule (Placebo Comparator): Placebo (capsules identically looking as acetazolamide capsules: 1 in the morning, 2 in the evening), orally. Medication starts 24 hours before ascent to 3200m until the morning after the second night at 3200m.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ACETAZOLAMIDE oral capsule — Administration of 125mg acetazolamide in the morning, 250mg in the evening, starting 24 hours before departure to 3200m
  Arms: ACETAZOLAMIDE oral capsule
Drug: Placebo oral capsule — Administration of equally looking placebo capsules in the morning and evening, starting 24 hours before departure to 3200m
  Arms: PLACEBO oral capsule

SUMMARY:
This trial will evaluate the effect of acetazolamide (375 mg per day) vs. placebo on right ventricular function during exercise at acute altitude exposure in patients with COPD.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind parallel trial evaluating the effect of acetazolamide (375 mg per day) vs. placebo on right ventricular function during exercise in lowlanders with chronic obstructive pulmonary disease travelling to altitude. Participants living in the Bishkek area, Kyrgyzstan (760m), will be transferred by car within 4h to the Tuja Ashu high altitude clinic (3200 m), and stay there for 2 days. Acetazolamide 375mg/day (or placebo) will be administered 24 hours before departure at 760 m and during the stay at altitude. Outcomes will be assessed during the stay at 3200 m.

Right ventricular function will be assessed during graded cycling on an ergometer by transthoracic echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, age 18-75 yrs.
* COPD diagnosed according to GOLD, FEV1 40-80% predicted, SpO2 ≥92% at 750 m.
* Born, raised and currently living at low altitude (<800m).
* Written informed consent.

Exclusion Criteria:

* COPD exacerbation, very severe COPD with hypoxemia at low altitude (FEV1/FVC <0.7, FEV1 <40% predicted, oxygen saturation on room air <92% at 750 m).
* Comorbidities such as uncontrolled cardiovascular disease, i.e., unstable systemic arterial hypertension, coronary artery disease; previous stroke; OSA; pneumothorax in the last 2 months.
* Internal, neurologic, rheumatologic or psychiatric disease including current heavy smoking (>20 cigarettes per day)
* Known renal failure or allergy to acetazolamide and other sulfonamides

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
pulmonary artery pressure during exercise | Day 2 at 3200m
  Difference in change of tricuspid pressure gradient during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer

SECONDARY OUTCOMES:
pulmonary artery pressure during exercise | Day 2 at 760 m and 3200 m
  Difference in altitude-induced change of tricuspid pressure gradient during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
cardiac output during exercise | Day 2 at 3200m
  Difference in change of cardiac output during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer
cardiac output during exercise | Day 2 at 760 m and 3200 m
  Difference in altitude-induced change of cardiac output during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
PAP/CO slope during exercise | Day 2 at 3200m
  Difference in change of PAP/CO slope during exercise between acetazolamide and placebo group at altitude, measured by transthoracic echocardiography during graded cycling on an ergometer
PAP/CO slope during exercise | Day 2 at 760 m and 3200 m
  Difference in altitude-induced change of PAP/CO slope during exercise between acetazolamide and placebo group, measured by transthoracic echocardiography during graded cycling on an ergometer
Oxygen saturation | Day 2 and 3200 m
  Difference in altitude-induced change during exercise of oxygen saturation between acetazolamide and placebo group, measured by pulse oximeter
Oxygen saturation | Day 2 at 760 m and 3200 m
  Difference in change of oxygen saturation during exercise between acetazolamide and placebo group, measured by pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, MD, Principal Investigator — University of Zurich; Talant M Sooronbaev, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided